CLINICAL TRIAL: NCT04544345
Title: Impact of Atrio-ventricular Optimization With His Bundle Pacing on Treatment of Atrio-ventricular Dromotropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Anja Zupan Mežnar, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMCLj-AVdromHis
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Atrioventricular Block; Atrioventricular Dyssynchrony
Keywords: AV block; His bundle pacing; AV dyssynchrony; AV optimization; AV dromotropathy; First degree AV block; Peak oxygen uptake
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- His bundle pacing, AV optimized (Experimental): Pacemaker programmed to DDD mode with ventricular lead placed on the bundle of His and echocardiographically optimized AV delay.
  Interventions: Device: His bundle pacing, AV optimized
- Backup VVI pacing (Sham Comparator): Pacemaker programmed to ventricular only pacing with low base rate (40/min) to allow intrinsic rhythm.
  Interventions: Device: Backup VVI pacing

INTERVENTIONS:
Device: His bundle pacing, AV optimized — A Select Secure 3830 (Medtronic, MN, USA) pacing lead will be placed on the bundle of His. In case of unsuccessful His capture, left bundle branch area pacing is going to be targeted. Pacemaker will be programmed to a low base rate and a high tracking rate to allow for intrinsic sinus rhythm. AV delay will be optimized with echocardiography to the shortest AV delay without truncation of the A wave on transmitral pulse wave doppler.
  Arms: His bundle pacing, AV optimized
Device: Backup VVI pacing — Pacemaker will be programmed to VVI (ventricular only) mode with low base rate as to allow for intrinsic sinus rhythm without AV optimization.
  Arms: Backup VVI pacing

SUMMARY:
This study aims to determine the clinical and hemodynamic benefit of atrio-ventricular (AV) resynchronization with His bundle pacing in patients with symptomatic first degree AV block.

DETAILED DESCRIPTION:
The term AV dyssynchrony was introduced by Salden F. and coauthors in 2018. It stands for the adverse effects of AV dyssynchrony due to PR interval prolongation. According to the ESC and ACC guidelines, severe first degree AV block is an IIa indication for permanent pacemaker implantation, yet data on these patients' clinical outcomes are scarce. To independently determine the impact of AV resynchronization, His bundle pacing will be used to avoid intraventricular desynchronization.

Symptomatic patients with severe first-degree AV block and echocardiographically proven AV dyssynchrony will be included in the study.

All patients will receive a dual-chamber pacemaker with an atrial lead positioned in the right atrium and ventricular lead placed on the bundle of His. In a single-blind cross-over design, patients will be randomized to AV sequential His bundle pacing with echo-guided AV optimization or back-up VVI pacing mode. Each study period will last for three months. At the end of both periods, cardiopulmonary exercise testing, complete echocardiographic study, and clinical evaluation will be performed.

Peak oxygen uptake and echocardiography-based hemodynamic parameters in both periods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* First OR second degree Mobitz type 1 atrioventricular block with a PR interval > 250 ms
* left ventricular ejection fraction > 50%
* echocardiographic criteria of atrioventricular dyssynchrony (diastolic filling time/RR interval ratio < 0,4 OR fusion of E and A waves OR diastolic mitral regurgitation)
* symptoms on exertion (dyspnea, palpitations)
* insufficient shortening of PR interval during exercise (PR interval > 200 ms at heart rate of 100 beats per minute)

Exclusion Criteria:

* left ventricular ejection fraction < 50%
* third degree atrioventricular block
* atrial fibrillation
* sinus node disease
* left bundle branch block
* right bundle branch block
* ventricular arrhythmia that indicates implantation of cardioverter defibrillator
* consumption of drugs that influence atrioventricular conduction
* active bacterial infection
* inability to undergo cardiopulmonary exercise test
* anaemia (haemoglobin concentration < 100 g/L)
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Changes in exercise capacity | Baseline, 3 months, 6 months
  Measured by peak oxygen consumption on cardiopulmonary exercise test
Changes in left ventricular stroke volume | Baseline, 3 months, 6 months
  Measured by echocardiography
Changes in quality of life using the 5 level EQ-5D questionnaire | Baseline, 3 months, 6 months
  EQ-5D is a standardized measure of health status consisting of 2 pages - the EQ-5D descriptive system (descriptive system with five levels) and the EQ visual analog scale ranging from 0 (worst state) to 100 (best state).

SECONDARY OUTCOMES:
Changes in left ventricular volume | Baseline, 3 months, 6 months
  End diastolic volume measured echocardiographicaly with biplane Simpson method
Changes in left atrial volume | Baseline, 3 months, 6 months
  Left atrial volume indexed by body surface area measured by echocardiography
Changes in the measure of left ventricular mechanical dyssynchrony | Baseline, 3 months, 6 months
  Measured by mid-ventricular radial speckle-tracking strain with an anteroseptal to posterior wall delay (AS-P delay)
Changes in QRS complex width | Baseline, 3 months, 6 months
  Measured by electrocardiogram
Changes in pacing thresholds | Baseline, 3 months, 6 months
  Measured during device check
Changes in sensing of R wave | Baseline, 3 months, 6 months
  Measured during device check
Changes in lead impedance | Baseline, 3 months, 6 months
  Measured during device check
Fluoroscopy time | Baseline
  Time of fluoroscopy use during device implantation
Adverse events | through study completion, an average of one year
  Any of the following adverse events: pocket hematoma, pneumothorax, hemothorax, cardiac tamponade, lead dislocation, lead perforation, cardiac implantable device infection

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Salden FCWM, Kutyifa V, Stockburger M, Prinzen FW, Vernooy K. Atrioventricular dromotropathy: evidence for a distinctive entity in heart failure with prolonged PR interval? Europace. 2018 Jul 1;20(7):1067-1077. doi: 10.1093/europace/eux207. PMID 29186415
- [Background] Aro AL, Anttonen O, Kerola T, Junttila MJ, Tikkanen JT, Rissanen HA, Reunanen A, Huikuri HV. Prognostic significance of prolonged PR interval in the general population. Eur Heart J. 2014 Jan;35(2):123-9. doi: 10.1093/eurheartj/eht176. Epub 2013 May 14. PMID 23677846
- [Background] Iliev II, Yamachika S, Muta K, Hayano M, Ishimatsu T, Nakao K, Komiya N, Hirata T, Ueyama C, Yano K. Preserving normal ventricular activation versus atrioventricular delay optimization during pacing: the role of intrinsic atrioventricular conduction and pacing rate. Pacing Clin Electrophysiol. 2000 Jan;23(1):74-83. doi: 10.1111/j.1540-8159.2000.tb00652.x. PMID 10666756
- [Background] European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE. 2013 ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Europace. 2013 Aug;15(8):1070-118. doi: 10.1093/europace/eut206. Epub 2013 Jun 24. No abstract available. PMID 23801827
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Kiehl EL, Makki T, Kumar R, Gumber D, Kwon DH, Rickard JW, Kanj M, Wazni OM, Saliba WI, Varma N, Wilkoff BL, Cantillon DJ. Incidence and predictors of right ventricular pacing-induced cardiomyopathy in patients with complete atrioventricular block and preserved left ventricular systolic function. Heart Rhythm. 2016 Dec;13(12):2272-2278. doi: 10.1016/j.hrthm.2016.09.027. PMID 27855853
- [Background] Sharma PS, Dandamudi G, Naperkowski A, Oren JW, Storm RH, Ellenbogen KA, Vijayaraman P. Permanent His-bundle pacing is feasible, safe, and superior to right ventricular pacing in routine clinical practice. Heart Rhythm. 2015 Feb;12(2):305-12. doi: 10.1016/j.hrthm.2014.10.021. Epub 2014 Oct 22. PMID 25446158
- [Background] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Background] Kutyifa V, Stockburger M, Daubert JP, Holmqvist F, Olshansky B, Schuger C, Klein H, Goldenberg I, Brenyo A, McNitt S, Merkely B, Zareba W, Moss AJ. PR interval identifies clinical response in patients with non-left bundle branch block: a Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy substudy. Circ Arrhythm Electrophysiol. 2014 Aug;7(4):645-51. doi: 10.1161/CIRCEP.113.001299. Epub 2014 Jun 24. PMID 24963007
- [Background] Joshi NP, Stopper MM, Li J, Beshai JF, Pavri BB. Impact of baseline PR interval on cardiac resynchronization therapy outcomes in patients with narrow QRS complexes: an analysis of the ReThinQ Trial. J Interv Card Electrophysiol. 2015 Aug;43(2):145-9. doi: 10.1007/s10840-015-9999-y. Epub 2015 Apr 29. PMID 25921348
- [Background] Zhang J, Guo J, Hou X, Wang Y, Qian Z, Li K, Ge P, Zou J. Comparison of the effects of selective and non-selective His bundle pacing on cardiac electrical and mechanical synchrony. Europace. 2018 Jun 1;20(6):1010-1017. doi: 10.1093/europace/eux120. PMID 28575215